CLINICAL TRIAL: NCT03401411
Title: Intensive Care Unit (ICU) Triage Practices in a Cancer Hospital
Brief Title: ICU Triage Practices in a Cancer Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2009-0450
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Intensive Care Units; Triage
Keywords: ICU; ICU Triage Practices; Cancer Patients; Oncology ICU
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard SCCMP (Experimental): Health care provider completes triage survey of 15 fictional patient case scenarios using the standard SCCMP to prioritize each for admission.
  Interventions: Behavioral: Survey
- SCCMP + Algorithm-based Triage Tool (Experimental): Health care provider completes triage survey of 15 fictional patient case scenarios using SCCMP in addition to a newly designed flowchart-based triage guide to prioritize each for admission.
  Interventions: Behavioral: Survey; Behavioral: Algorithm-based Triage Tool

INTERVENTIONS:
Behavioral: Survey — Survey of 15 fictional patient case scenarios to be assessed by participant using the standard prioritization or modified SCCMP to prioritize each patient scenario into one of a 5-point likert-scale categories for ICU admission. SCCMP scale categorized as 1-Critically ill to 4-Less likely to require ICU.
  Other Names: Society of Critical Care Medicine Prioritization Model
Behavioral: Algorithm-based Triage Tool — Newly designed flowchart-based triage guide to prioritize each patient case scenario into one of the 5-point likert-scale categories, used in conjunction with SCCMP for ICU admission.
  Arms: SCCMP + Algorithm-based Triage Tool

SUMMARY:
The primary objective of this study is aimed at analyzing the ICU triage practices of clinicians at a cancer hospital with and without the use of an algorithm-based triage tool, and to assess whether or not the triage tool improves the consensus amongst practioners on the prioritization of patients for ICU admission. Secondary objectives include assessment of whether or not triage practices based on guidelines correlate with what is done in actual practice.

DETAILED DESCRIPTION:
This is a prospective study designed to evaluate the ICU triage practices of clinicians at MD Anderson Cancer Center using the standard Society of Critical Care Medicine Prioritization Model (SCCMP) versus a uniquely designed flowchart-based triage tool created specifically for the oncologic setting.

Study participants will initially receive either an email explaining the study and asking if they would agree to participate in the survey, or a hard copy of an identical letter. Their participation will remain anonymous, and will strictly be on a volunteer basis. If the participant wishes to participate, they will be given either a link to the survey using an institutionally improved electronic survey tool, or alternatively a hard copy of the survey with identical instructions.

The survey consists of 15 fictional patient case scenarios, and participants will be asked to use the modified SCCMP to prioritize each patient scenario into one of the 5-point likert-scale categories for admission. The participants will be randomized with 1:1 ratio to use either a) the standard SCCMP or b) the SCCMP in addition to a newly designed flowchart-based triage guide to prioritize each patient case scenario into one of the 5-point likert-scale categories.

ELIGIBILITY:
Inclusion Criteria:

1) Study participant must be a health care provider who frequently refers or accepts oncologic patients to the ICU

Exclusion Criteria:

1) none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Agreement among clinicians for each of triage tools: SCCMP Standard versus SCCMP + Algorithm-based Triage Tool | 20 minutes for participant survey completion
  Survey responses used to evaluate the ICU triage practices of clinicians using the standard SCCMP versus a uniquely designed flowchart-based triage tool created specifically for the oncologic setting. Participants are randomized to use either a) the standard SCCMP or b) the SCCMP in addition to a newly designed flowchart-based triage guide to prioritize 15 fictional patient case scenarios into one of the 5-point likert-scale categories for admission.
  SCCMP system defines those that will benefit most from the ICU (Priority 1) to those that will not benefit at all (Priority 4) from ICU admission. Reported proportion of clinicians choosing category i in the 5-point likert-scale, i=1, 2, 3, 4a or 4b, for a particular patient case. The range of the entropy is between 0 (perfect agreement among the clinicians) and 1.61 (total disagreement among the clinicians).

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Rathi, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (3):
- United States (2):
  - Latino-American Critical Care Trial Network (LACTIN), Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- 5th International Oncology Course Conference, Manta, Manabí Province, Ecuador

REFERENCES:
- See also: The University of Texas (UT) MD Anderson Cancer Center Official Website — http://www.mdanderson.org